CLINICAL TRIAL: NCT04342598
Title: Case Control Study of Vitamin D Status and Adult Multidrug-resistant Pulmonary Tuberculosis in Maharashtra, India
Status: Completed | Type: Observational
Sponsor: Harvard School of Public Health (HSPH) (Other)
Collaborators: Foundation for Medical Research (Other); Municipal Corporation of Greater Mumbai, India (Unknown)
Responsible Party: Principal Investigator, Wafaie Fawzi, Professor of Nutrition, Epidemiology, and Global Health, Harvard School of Public Health (HSPH)
Other Study IDs: IRB19-0237
Record Dates: First submitted 2020-04-07; First posted 2020-04-13 (Actual); Last update posted 2021-02-25 (Actual); Status verified 2021-02

CONDITIONS: Multi-drug Resistant Tuberculosis
Keywords: Multi-drug resistant tuberculosis; Extensively drug-resistant tuberculosis; Vitamin D; Vitamin D deficiency; Tuberculosis; Latent tuberculosis infection; Diet
MeSH Terms: conditions — Tuberculosis, Multidrug-Resistant; Extensively Drug-Resistant Tuberculosis; Vitamin D Deficiency; Tuberculosis; Latent Tuberculosis | interventions — Diet

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Adult outpatient pulmonary MDR-TB patients
  Interventions: Other: Serum Vitamin D
- Household contact controls
  Interventions: Other: Serum Vitamin D
- Non-household contact controls
  Interventions: Other: Serum Vitamin D

INTERVENTIONS:
Other: Serum Vitamin D — Primary exposure assessed will be serum vitamin D (25(OH)D). Diet will also be assessed via Food Frequency Questionnaire.
  Other Names: Diet

SUMMARY:
India has the highest incidence of and mortality from multi-drug resistant tuberculosis (MDR-TB) globally. Vitamin D status may be an important determinant of MDR-TB infection and treatment outcomes; however, observational evidence is insufficient to support its use as an adjunct therapy or prophylaxis. Using a case-control design, this study will evaluate the relationship between vitamin D status and active MDR-TB disease among adult outpatient pulmonary MDR-TB cases, household contact controls, and matched controls from the general population (non-household controls) in Mumbai, India. This study will also evaluate the cross-sectional association between vitamin D status and TB infection among household contact controls and non-household controls, and collect formative data in preparation for future randomized controlled trials of vitamin D in MDR-TB prevention and treatment in India.

DETAILED DESCRIPTION:
To combat the substantial global burdens of TB and MDR-TB, novel treatment strategies and expanded prevention efforts are critical. Although vitamin D supplementation shows promise in both of these areas, additional observational evidence is needed to support future randomized clinical trials. This case-control study in Mumbai, India will clarify associations between vitamin D status, active MDR-TB disease and TB infection to expand the evidence-base and inform the design of future trials of vitamin D supplementation for use in MDR-TB infection. This study will assess vitamin D status, diet, and anthropometry among adult outpatient MDR-TB cases and controls in Mumbai, India and assess TB infection among controls. The specific aims are: 1) evaluate the association between vitamin D status and active MDR-TB infection; 2) evaluate the association between vitamin D status and TB infection among controls; 3) collect formative data to inform the design of future randomized clinical trials evaluating vitamin D supplementation and other interventions in MDR-TB treatment and prevention. To fulfill the first aim, a case-control study will be conducted comparing vitamin D status between pulmonary MDR-TB cases (including extensively drug-resistant (XDR) and pre-XDR cases) and two sets of controls: 1) household controls (recruited from the cases' household contacts) and 2) non-household controls (recruited from non-respiratory departments of local hospitals). The second aim will involve a cross-sectional study among controls assessing the association between vitamin D status and TB infection using QuantiFERON-TB (QFT-TB) interferon-gamma release assays.

ELIGIBILITY:
1. Inclusion criteria for cases:

   * Currently receiving outpatient treatment for MDR-TB according to standard of care (including new cases and those who have been on treatment for no more than one month)
   * Residence in Mumbai M/E, M/W or H/E ward for at least six months
   * 18-60 years old
   * Permanently living with at least two eligible controls
   * Confirmation that they have disclosed their TB status to household and will allow inclusion of their household members in the study
2. Inclusion criteria for household contact controls:

   * Was a permanent member of the index case's household for at least one year prior to the case's DR TB diagnosis
   * No symptoms of active TB disease
   * Residence in Mumbai M/E, M/W or H/E ward for at least six months
   * 18-60 years old
3. Inclusion criteria for non-household controls:

   * 18 - 60 years of age
   * Residence in Mumbai M/E, M/W or H/E ward for at least six months
   * No symptoms of active TB disease
   * No history of household contact with a TB patient in last 2 years

Exclusion criterion for both cases and controls:

• Pregnancy.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Adult pulmonary outpatient MDR-TB cases, household contact controls and non-household controls residing in Mumbai in Maharashtra state, India
Sampling Method: Non-Probability Sample
Enrollment: 352 (Actual)
Dates: Start 2020-01-27 (Actual); Primary Completion 2020-12-17 (Actual); Study Completion 2020-12-17 (Actual)

PRIMARY OUTCOMES:
Adult pulmonary multi-drug resistant tuberculosis | Baseline
  Defined by the Guidelines on Programmatic Management of Drug-Resistant TB in India. Includes cases with MDR-TB (resistant to both isoniazid and rifampicin with or without resistance to other first-line drugs), pre-XDR-TB(MDR-TB patients with additional resistance to any/all fluoroquinolones or any/all second-line drugs, or XDR-TB (MDR-TB patients who are additionally resistant to at least one fluoroquinolone and a second-line drug).

SECONDARY OUTCOMES:
Latent TB infection among controls | Baseline
  Assessed using QuantiFERON-TB (QFT-TB) interferon-gamma release assays.

CONTACTS AND LOCATIONS:
Overall Officials: Wafaie W Fawzi, MBBS, MPH, MS, DrPH, Principal Investigator — Harvard School of Public Health (HSPH)
Locations (1):
- Foundations for Medical Research, Mumbai, Maharashtra, India

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Digvijaya, Mittal S, Mittal P, Singh R, Gupta S, Singh T, Khan R, Alzobaidi N, Alhalmi A. Vitamin D Fortification: A Promising Approach to Overcome Drug Resistance and Tolerance in Therapeutic Interventions. Scientifica (Cairo). 2024 Nov 22;2024:9978076. doi: 10.1155/2024/9978076. eCollection 2024. PMID 39618688
- [Derived] Mistry N, Hemler EC, Dholakia Y, Bromage S, Shukla A, Dev P, Govekar L, Tipre P, Shah D, Keshavjee SA, Fawzi WW. Protocol for a case-control study of vitamin D status, adult multidrug-resistant tuberculosis disease and tuberculosis infection in Mumbai, India. BMJ Open. 2020 Nov 12;10(11):e039935. doi: 10.1136/bmjopen-2020-039935. PMID 33184081